CLINICAL TRIAL: NCT06949111
Title: Efficacy and Safety of Conversion Therapy for pMMR/MSS T4M0 Colon Cancer Patients Treated With Radiotherapy and Systemic Therapy: a Prospective, Open-label, Multi-center, Randomized Controlled Trial（Neo-Color）
Brief Title: Radiotherapy + Systemic Therapy as Conversion Therapy for pMMR/MSS T4M0 Colon Cancer（Neo-Color）
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025044
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer
Keywords: Locally advanced colon cancer; Neoadjuvant chemoradiotherapy; Immune checkpoint inhibitors; Complete response rate; Radiotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Radiotherapy; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy + Systemic Therapy (Experimental): Patients undergo radiotherapy (36-41.4 Gy/20-23f). Concurrently, patients will receive Capecitabine (825 mg/m², bid, on radiotherapy days). At 23.4 Gy/13f of radiotherapy, patients will be administered Iparomlimab-Tuvonralimab (5 mg/kg) for one cycle. 1-2 weeks after completing the 36-41.4 Gy radiotherapy, patients will begin 4 cycles of CAPOX plus Iparomlimab-Tuvonralimab (5 mg/kg).
  All patients were evaluated for therapeutic efficacy 2-3 weeks after above therapy. Patients met the criteria for complete remission (cCR) could choose either surgery or not. For patients who chose surgery, four cycles of CAPOX were administered 4-6 weeks after surgery. For patients who did not choose surgery, 4 cycles of CAPOX was continued.
  For patients did not meet the cCR criteria, surgery and 4 cycles of CAPOX was recommended. Patients who refused surgery continued to receive 4 cycles of CAPOX. If the second response evaluation met the cCR criteria, patients were included in the primary end point.
  Interventions: Radiation: radiotherapy; Drug: CAPOX; Drug: Capecitabine; Drug: Iparomlimab and Tuvonralimab Injection
- Chemotherapy Alone (Active Comparator): Patients will receive 4 cycles of CAPOX. Then all patients were evaluated for therapeutic efficacy 2-3 weeks after therapy. Patients met the criteria for complete remission (cCR) could choose either surgery or not. For patients who chose surgery, four cycles of CAPOX were administered 4-6 weeks after surgery. For patients who did not choose surgery, 4 cycles of CAPOX was continued.
  For patients did not meet the cCR criteria, surgery and 4 cycles of CAPOX was recommended. Patients who refused surgery continued to receive 4 cycles of CAPOX. If the second response evaluation met the cCR criteria, patients were included in the primary end point.
  Interventions: Drug: CAPOX

INTERVENTIONS:
Radiation: radiotherapy — Radiotherapy: Administer three-dimensional conformal/intensity-modulated/TOMO radiotherapy with a conventional fractionation schedule of 36-41.4 Gy in 20-23 fractions (1.8 Gy per fraction).
  Arms: Radiotherapy + Systemic Therapy
Drug: CAPOX — 4 cycles, Oxaliplatin 130 mg/m², Capecitabine 825 mg/m²
Drug: Capecitabine — Administer Capecitabine at a dose of 825 mg/m², twice daily, orally on radiotherapy days
  Arms: Radiotherapy + Systemic Therapy
Drug: Iparomlimab and Tuvonralimab Injection — IV, 5 mg/kg every 3 weeks
  Arms: Radiotherapy + Systemic Therapy

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of conversion therapy using radiotherapy combined with systemic treatment (chemotherapy + immune checkpoint inhibitors) for patients with pMMR/MSS T4M0 stage colon cancer. The main questions it aims to answer are:

1. Can the combination of radiotherapy and systemic treatment improve the R0 resection rate and complete response (CR) rate compared to chemotherapy alone?
2. Does this combination therapy enhance the tumor immune microenvironment, leading to better long-term outcomes?

Researchers will compare the experimental group receiving concurrent chemoradiotherapy (CCRT) followed by 4 cycles of CAPOX + Iparomlimab and Tuvonralimab Injection with the control group receiving 4 cycles of CAPOX alone to see if the combination therapy offers superior efficacy.

Participants will:

1. Undergo preoperative CCRT combined with one cycle of Iparomlimab and Tuvonralimab Injection, followed by 4 cycles of CAPOX + Iparomlimab and Tuvonralimab Injection in the experimental group.
2. Receive 4 cycles of CAPOX in the control group.
3. After the initial treatment regimen, surgical candidates will undergo surgery followed by an additional 4 cycles of CAPOX. Non-surgical candidates will continue with 4 more cycles of CAPOX, completing a total of 8 cycles. Efficacy will be re-evaluated after the completion of 8 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, no restriction on gender.
2. ECOG performance status of 0-1.
3. Histopathologically confirmed diagnosis of colon adenocarcinoma (including mucinous adenocarcinoma), identified as pMMR/MSS type; the primary tumor site must be specified (left colon defined as from the splenic flexure to the rectosigmoid junction, right colon defined as from the cecum to the proximal splenic flexure).
4. Baseline imaging (enhanced CT/MRI) confirms clinical staging as cT4NanyM0 according to the AJCC 8th edition staging criteria.
5. Laboratory criteria prior to enrollment must meet the following ranges:

(1) Hematology: Absolute neutrophil count ≥ 1.5 × 10^9/L, platelets ≥ 100 × 10^9/L, hemoglobin ≥ 90 g/L.

(2) Liver and renal function: ALT/AST ≤ 2.5 × ULN, total bilirubin ≤ 1.5 × ULN, creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 mL/min (Cockcroft-Gault formula).

(3) Coagulation function: INR ≤ 1.5, APTT ≤ 1.5 × ULN (for those not on anticoagulation therapy).

6.Women of childbearing potential and men must agree to use effective contraception during the study and for 6 months after the last treatment.

7.Willingness to sign a written informed consent form and commit to completing the entire treatment and follow-up plan.

Exclusion Criteria:

1. Histological type of neuroendocrine carcinoma, squamous cell carcinoma, or other non-adenocarcinoma components comprising more than 50%.
2. Presence of distant metastasis (including peritoneal metastasis, non-regional lymph node metastasis, or organ metastasis).
3. Previous radiotherapy, chemotherapy, targeted therapy, or immunotherapy for colon cancer.
4. Active autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis requiring long-term immunosuppressive therapy).
5. Active infections (e.g., HIV, positive HBV/HCV viral load requiring antiviral treatment for stabilization).
6. Severe cardiovascular diseases (e.g., myocardial infarction within 6 months, unstable angina, uncontrolled hypertension >160/100 mmHg).
7. History of other malignancies (except for cured non-melanoma skin cancer, cervical carcinoma in situ, etc., with a disease-free period of ≥5 years).
8. Uncontrolled diabetes (HbA1c > 8%) or thyroid dysfunction (TSH outside the normal range requiring medication).
9. Severe chronic bowel diseases (e.g., active Crohn's disease, ulcerative colitis).
10. History of radiation enteritis or extensive abdominal adhesions affecting radiotherapy target delineation.
11. Unrecovered bone marrow suppression (ANC < 1.5 × 10^9/L, PLT < 100 × 10^9/L, Hb < 90 g/L).
12. Liver function with Child-Pugh score ≥ B or renal function with eGFR < 60 mL/min/1.73 m².
13. Pregnant or breastfeeding women (blood/urine HCG test required during screening).
14. Cognitive impairment or history of psychiatric disorders affecting treatment compliance.
15. Concurrent participation in other interventional clinical trials.
16. Patients deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Tumor Complete Response (CR) Rate | 2 years
  CR including pCR and cCR

SECONDARY OUTCOMES:
MPR rate | 4 years
R0 Resection Rate | 4 years
Adjacent Organ Preservation Rate | 4 years
EFS rate | 3 years
OS rate | 3 years
Adverse events | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- the Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided